CLINICAL TRIAL: NCT04156230
Title: A Phase 2, Open-label, Non-randomized, Single Center Study to Assess Diagnostic Validity of [18F]GP1 Positron Emission Tomography/Computed Tomography for Acute Deep Vein Thrombosis of the Lower Extremities in Symptomatic Patients
Brief Title: Diagnostic Validity of [18F]GP1 PET for Diagnosing Acute Deep Vein Thrombosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dae Hyuk Moon (Other)
Responsible Party: Sponsor-Investigator, Dae Hyuk Moon, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GP1-1901
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Venous Thrombosis
Keywords: Positron-Emission Tomography; Ultrasonography; Platelet Activation; Data Accuracy
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Symptomatic subjects with a pretest score of deep vein thrombosis likely (Wells score ≥ 2) or a positive D-dimer test will receive [18F]GP1 PET/CT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Deep vein thrombosis (Experimental): Subjects with Deep vein thrombosis will receive a single IV injection of [18F] GP1
  Interventions: Drug: [18F]GP1 positron emission tomography/computed tomography

INTERVENTIONS:
Drug: [18F]GP1 positron emission tomography/computed tomography — A radioactive dose of 250 MBq of the study drug with a total quantity of ≤ 10 µg will be administered as slow intravenous bolus injection over up to 60 seconds. PET/CT examinations will be performed at 120 ± 15 min after the administration of [18F]GP1.

SUMMARY:
The first-in-human study of [18F]GP1 positron emission tomography/computed tomography (PET/CT) showed that [18F]GP1 is safe and promising novel PET tracer for imaging acute venous thromboembolism with favorable biodistribution and pharmacokinetics in patients. The goal of this phase 2 study is to evaluate whether [18F]GP1 PET/CT is sensitive and specific for the diagnosis of acute deep vein thrombosis in the appropriate patient population and clinical setting. This study will provide preliminary evidence of efficacy and expand the safety database in a larger group of patients who were suspected of having acute deep vein thrombosis. This study will further optimize image acquisition techniques, and develop methods and criteria by which [18F]GP1 PET/CT will be evaluated. Other critical questions about [18F]GP1 biodistribution including [18F]GP1 uptake in pulmonary and systemic arteries will be evaluated.

DETAILED DESCRIPTION:
This study is an open label, non-randomized, single center, intervention study. An estimated 63 symptomatic subjects with a pretest score of deep vein thrombosis likely (Wells score ≥ 2) or a positive D-dimer test will receive [18F]GP1 PET/CT to evaluate the diagnostic validity of [18F]GP1 PET/CT for detecting deep vein thrombosis foci in lower extremities.

The study comprises 3 periods: screening, treatment, and follow-up. The screening period starts with the patient's signature on the informed consent form and ends with assignment to treatment that is inclusion of the subject for treatment. The treatment period starts with baseline measurements, and ends with the last measurement/procedure on the day of intravenous injection of 250 MBq of [18F]GP1. The follow-up period contains the end-of-study interview. Key measurement is the PET/CT image acquisition about 120 minutes after the single injection of [18F]GP1 This study includes venous ultrasonography of deep vein thrombosis as a valid reference standard. [18F]GP1 PET/CT will be assessed qualitatively and quantitatively by three experienced readers.

This study will be monitored regularly by a clinical research associate from the sponsor or a designated contract research organization. Data quality and study integrity will be assessed. The investigator will document the items that are required to evaluate the study in the subject files. Data required according to this protocol are to be recorded on the case report forms provided by the sponsor as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be enrolled if he/she meets all of the following inclusion criteria.

  * Subject is aged between 19 and 79 years and male or female of any race/ethnicity.
  * Patient has a first episode of clinically suspected acute deep vein thrombosis of the lower extremity within 14 days prior to the planned [18F]GP1 PET/CT.
  * The pretest probability for deep vein thrombosis is likely by two-level Wells score (≥ 2), or the D-dimer test is positive.
  * Subject underwent or is scheduled to undergo venous ultrasonography within 7 days of [18F]GP1 PET/CT:
  * Patient has Eastern Cooperative Oncology Group performance status of 0-2 at time of screening.

Exclusion Criteria:

* A subject is to be excluded from the study if he/she does not fulfill the inclusion criteria or display any of the following criteria.

  * Subject or subject's legally acceptable representative does not provide written informed consent.
  * Subject has a previous history of objectively diagnosed deep vein thrombosis or pulmonary embolism.
  * Subject has symptoms of acute deep vein thrombosis lasting for longer than 4 weeks at time of screening.
  * Subject is suspected to have pulmonary embolism with shock or hypotension
  * Subject had pretreatment with glycoprotein IIb/IIIa inhibitors within 15 days before the administration of [18F]GP1.
  * Anticancer chemotherapy is scheduled to be given to subject before or within 24 hours after administration of [18F]GP1.
  * Female subject is pregnant or nursing. Exclusion of the possibility of pregnancy is made by one of the following: 1) woman is physiologically post-menopausal (cessation of menses for more than 2 years), or 2) woman is surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy). If the woman is of childbearing potential, a urine pregnancy test performed within 24 hours immediately prior to administration of [18F]GP1 has to be negative and the women is advised to apply contraceptive measures during her participation in this study.
  * Subject has concurrent severe and/or uncontrolled and/or unstable medical disease other than cancer (e.g. congestive heart failure, acute myocardial infarction, severe pulmonary disease, chronic renal or hepatic disease) which could compromise participation in the study in the judgment of the investigator.
  * Subject is a relative of the investigator, student of the investigator or otherwise dependent.
  * Subject has been involved in another investigative clinical study involving administration of an investigational drug from preceding 4 weeks prior to the study enrollment or within 24 hours after administration of [18F]GP1.
  * Subject has been previously included in this study.
  * Subject has any other condition or personal circumstances that, in the judgment of the investigator, might make collection of complete data difficult or impossible.
  * Additive-related precautions: This investigational product contains sodium bisulfite, a sulfite that may cause allergic-type reactions including anaphylactic symptoms and life-threatening or less severe asthmatic episodes in certain susceptible people. The overall prevalence of sulfite sensitivity in the general population is unknown and probably low. Sulfite sensitivity is seen more frequently in asthmatic than in nonasthmatic people.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of qualitative [18F]GP1 PET/CT interpretation for the diagnosis of patients with acute proximal deep vein thrombosis | within 7 days of [18F]GP1 PET/CT
  Sensitivity = (the number of [18F]GP1 PET/CT-positive patients divided by the number of ultrasonography-positive patients) x 100; specificity = (the number of [18F]GP1 PET/CT-negative patients divided by the number of ultrasonography-negative patients) x 100.

SECONDARY OUTCOMES:
Area under the receiver operating characteristic curve, sensitivity and specificity of quantitative [18F]GP1 PET/CT interpretation for the diagnosis of patients with acute proximal deep vein thrombosis | Within 7 days of [18F]GP1 PET/CT
  Area under the receiver operating characteristic curve. Sensitivity = (the number of [18F]GP1 PET/CT-positive patients divided by the number of ultrasonography-positive patients) x 100; specificity = (the number of [18F]GP1 PET/CT-negative patients divided by the number of ultrasonography-negative patients) x 100.
Positive and negative percent agreement between qualitative [18F]GP1 PET/CT and ultrasonography interpretation for the diagnosis of patients with acute distal deep vein thrombosis | Within 7 days of [18F]GP1 PET/CT
  Positive percent agreement = (the number of [18F]GP1 PET/CT-positive patients divided by the number of ultrasonography-positive patients) x 100; negative percent agreement = (the number of [18F]GP1 PET/CT-negative patients divided by the number of ultrasonography-negative patients) x 100
Positive and negative percent agreement between quantitative [18F]GP1 PET/CT and ultrasonography interpretation for the diagnosis of patients with acute distal deep vein thrombosis | Within 7 days of [18F]GP1 PET/CT
  Positive percent agreement = (the number of [18F]GP1 PET/CT-positive patients divided by the number of ultrasonography-positive patients) x 100; negative percent agreement = (the number of [18F]GP1 PET/CT-negative patients divided by the number of ultrasonography-negative patients) x 100
Intra- and inter-reader variability of qualitative [18F]GP1 PET/CT interpretation for the assessment of acute proximal and distal deep vein thrombosis | Within 1 day of [18F]GP1 PET/CT
  kappa statistic
Detection rate of pulmonary embolism with [18F]GP1 PET/CT | Within 1 day of [18F]GP1 PET/CT
  The number of [18F]GP1 PET/CT-positive patients divided by the number of ultrasonography-positive patients) x 100; negative percent agreement = (the number of all patients who underwent [18F]GP1 PET/CT
Percent fraction of unmetabolized [18F]GP1 in plasma | Within 1 day of [18F]GP1 PET/CT
  Percentage
Incidence of treatment emergent adverse events | From the administration of [18F]GP1 to one day after [18F]GP1 PET/CT
  Number of participants with treatment emergent adverse events graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0)
Blood pressure | Pre-treatment and three hours after the administration of [18F]GP1
  mmHg
Heart rate | Pre-treatment and three hours after the administration of [18F]GP1
  beats/minute
Body temperature | Pre-treatment and three hours after the administration of [18F]GP1
  Celsius
Physical examination | Pre-treatment and three hours after the administration of [18F]GP1
  The limited physical examination will comprise: general appearance, skin, neck, lungs, heart, abdomen, and a limited neurological examination (mental status, motor strength and sensor perception).
Blood tests for safety | Pre-treatment and three hours after the administration of [18F]GP1
  The clinical laboratory safety parameters to be assessed are as follows: glutamate pyruvate transaminase, glutamate-oxaloacetate transaminase, alkaline phosphatase, total bilirubin, creatinine, potassium, sodium, total protein, blood urea nitrogen, albumin.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyuk Moon, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lohrke J, Siebeneicher H, Berger M, Reinhardt M, Berndt M, Mueller A, Zerna M, Koglin N, Oden F, Bauser M, Friebe M, Dinkelborg LM, Huetter J, Stephens AW. 18F-GP1, a Novel PET Tracer Designed for High-Sensitivity, Low-Background Detection of Thrombi. J Nucl Med. 2017 Jul;58(7):1094-1099. doi: 10.2967/jnumed.116.188896. Epub 2017 Mar 16. PMID 28302764
- [Background] Kim C, Lee JS, Han Y, Chae SY, Jin S, Sung C, Son HJ, Oh SJ, Lee SJ, Oh JS, Cho YP, Kwon TW, Lee DH, Jang S, Kim B, Koglin N, Berndt M, Stephens AW, Moon DH. Glycoprotein IIb/IIIa receptor imaging with 18F-GP1 positron emission tomography for acute venous thromboembolism: an open-label, non-randomized, first-in-human phase 1 study. J Nucl Med. 2018 Jun 29;60(2):244-9. doi: 10.2967/jnumed.118.212084. Online ahead of print. PMID 29959214
- [Background] Chae SY, Kwon TW, Jin S, Kwon SU, Sung C, Oh SJ, Lee SJ, Oh JS, Han Y, Cho YP, Lee N, Kim JY, Koglin N, Berndt M, Stephens AW, Moon DH. A phase 1, first-in-human study of 18F-GP1 positron emission tomography for imaging acute arterial thrombosis. EJNMMI Res. 2019 Jan 7;9(1):3. doi: 10.1186/s13550-018-0471-8. PMID 30617563
- [Background] Lee N, Oh I, Chae SY, Jin S, Oh SJ, Lee SJ, Koglin N, Berndt M, Stephens AW, Oh JS, Moon DH. Radiation dosimetry of [18F]GP1 for imaging activated glycoprotein IIb/IIIa receptors with positron emission tomography in patients with acute thromboembolism. Nucl Med Biol. 2019 May-Jun;72-73:45-48. doi: 10.1016/j.nucmedbio.2019.07.003. Epub 2019 Jul 10. PMID 31330411